CLINICAL TRIAL: NCT03866343
Title: Restriction of Dietary AGEs to Prevent Diabetes in Overweight Individuals: a Randomized Controlled Trial
Brief Title: Restriction of Dietary AGEs to Prevent Diabetes in Overweight Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL63215.068.17
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Advanced Glycation Endproducts; AGEs; Diet; Insulin Sensitivity/Resistance; Beta-cell Function; Vascular Function
MeSH Terms: conditions — Insulin Resistance | interventions — Glycation End Products, Advanced

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low AGE diet (Active Comparator): Subjects will be asked to consume a diet containing a low AGE content for 4 weeks.
  Interventions: Other: Diet low or high in advanced glycation endproducts
- High AGE diet (Other): Subjects will be asked to consume a diet containing a high AGE content for 4 weeks.
  Interventions: Other: Diet low or high in advanced glycation endproducts

INTERVENTIONS:
Other: Diet low or high in advanced glycation endproducts — All subjects will undergo an intervention consisting of a prescribed diet containing either a low or high quantity of AGEs during 4 continuous weeks.

SUMMARY:
Current efforts to arrest the epidemic of type 2 diabetes mellitus (T2DM) have had limited success. Thus there is an urgent need for effective approaches to prevent the development of T2DM. It is widely accepted that the current epidemic is driven by an increase in global food abundance and reduced food quality, making changes in diet a key determinant of the T2DM epidemic. Dietary factors can affect cardio-metabolic health; among these factors, advanced glycation end-products (AGEs) in food are potential risk factors for insulin resistance and T2DM.

AGEs are a heterogeneous group of unavoidable stable bioactive compounds. Endogenous formation of AGEs is a continuous naturally occurring process, and is the result of normal metabolism. However, increased formation of AGEs occurs during ageing and under hyperglycaemic conditions. AGEs are implicated in the development of diabetes and vascular complications.

Over the past several decades, methods of food processing have changed and meals now contain excess fat and sugar and are most susceptible for the formation of AGEs. In addition, AGEs in food are highly desirable due to their profound effect on shelf life, sterility, flavour, colour, and thus food consumption. Hence, a substantial portion of AGEs are derived from exogenous sources, particularly food. These exogenous AGEs are potential risk factors for insulin resistance and the development of T2DM. The investigators recently found that dietary AGEs represent a significant source of circulating AGEs, and have similar pathogenic properties compared to their endogenous counterparts including the development of insulin resistance and T2DM. Taken together, dietary AGEs are proposed to play a pivotal role in the development and progression of T2DM and its complications. Reduction of dietary intake of AGEs may therefore be an alternative strategy to reduce the risk of vascular disease and insulin resistance. The investigators therefore hypothesize that dietary restriction of AGEs in overweight individuals improves insulin sensitivity, β-cell function, and vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal obesity: waist circumference for men ≥ 102 cm, and for women ≥ 88 cm.
* Aged 18 years and older
* Caucasian (because of skin fluorescence and capillary microscopy measurements)

Exclusion Criteria:

* Diabetes (i.e. using anti-diabetic medication, fasting glucose >7.0 mmol/L, HbA1c >6.5%).
* Active or history of cardiovascular disease (e.g. stroke, coronary artery disease, peripheral vascular disease, congestive heart failure, cardiac shunts, cardiac surgery, pulmonary hypertension, cardiac arrhythmias, family history of cardiac arrhythmias or sudden cardiac death)
* Hyperlipidemia (defined as serum total cholesterol > 8 mmol/L or TG > 4 mmol/L)
* Lipid lowering medication (e.g. statins)
* Use of medication known to influence glucose metabolism, vascular function and/or lipid metabolism (e.g. statins, glucocorticosteroids, NSAID's)
* Inability to stop antihypertensive medication for 13 weeks. Exclusion of higher grade hypertension (> 179 mmHg SBP and/or > 109 mmHg DBP) in order not to expose subjects to unnecessary risks)
* Pulmonary or inflammatory disease
* Kidney failure or electrolyte disorders
* Pregnancy or lactation
* No change in use of oral anticonceptiva or IUD (12 weeks prior of during the intervention)
* Known allergic reaction to ultrasound contrast-agent
* Smoking (active or cessation <1 year prior to screening date).
* High alcohol usage (>4 U/day) or drug abuse
* Use of dietary supplements or an investigation product within the previous month
* Significant food allergies/intolerance
* Vegetarianism
* Subjects who intend to donate blood during the intervention or subjects who have donated blood less than three months before the start of the intervention.
* Participation in another biomedical trial during the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Difference after 4 weeks of intervention
  Assessed by hyperinsulinaemic-euglycaemic clamp

SECONDARY OUTCOMES:
Microvascular function | Difference after 4 weeks of intervention
  Assessed by contrast-enhanced ultrasound (CEUS) in skeletal muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Linkens AM, Houben AJ, Niessen PM, Wijckmans NE, de Goei EE, Van den Eynde MD, Scheijen JL, van den Waarenburg MP, Mari A, Berendschot TT, Streese L, Hanssen H, van Dongen MC, van Gool CC, Stehouwer CD, Eussen SJ, Schalkwijk CG. A 4-week high-AGE diet does not impair glucose metabolism and vascular function in obese individuals. JCI Insight. 2022 Mar 22;7(6):e156950. doi: 10.1172/jci.insight.156950. PMID 35133989